CLINICAL TRIAL: NCT01398644
Title: Erythrocytapheresis Versus Phlebotomy as Maintenance Therapy in Patients With Hereditary Hemochromatosis; a Randomised, Single Blinded Sequential, Cross-over Trial
Brief Title: Erythrocytapheresis Versus Phlebotomy as Maintenance Therapy in Hereditary Hemochromatosis (HH) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Maastricht University Medical Center (Other); Atrium Medical Center (Other); Radboud University Medical Center (Other); Orbis Medical Centre (Other)
Responsible Party: Principal Investigator, Eva Rombout, Transfusion specialist, Sanquin Research & Blood Bank Divisions
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 07-2-104
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Hereditary Hemochromatosis
Keywords: Phlebotomy; Therapeutic erythrocytapheresis; Hereditary Hemochromatosis; maintenance therapy
MeSH Terms: conditions — Hemochromatosis | interventions — Phlebotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phlebotomy -intervention phlebotomy (Active Comparator): Patients are treated with phlebotomy if ferritin level >50 ug/l
  Interventions: Other: Phlebotomy and erythrocytapheresis
- Erythrocytapheresis (Experimental): Patients are treated with erythrocytapheresis if serum ferritin level >50ug/l
  Interventions: Other: Phlebotomy and erythrocytapheresis

INTERVENTIONS:
Other: Phlebotomy and erythrocytapheresis — Phlebotomy- removal of 500 ml whole blood Erythrocytapheresis- removal of 300-800 ml erythrocytes

SUMMARY:
Hereditary hemochromatosis (HH) is a genetic disorder of iron metabolism, resulting in excessive iron overload. Phlebotomy is currently the standard therapy. More recently Therapeutic Erythrocytapheresis (TE) has become a new therapeutic modality, which potentially offers a more efficient method to remove iron overload with fewer procedures.In the proposed clinical trial the investigators will examine whether TE can keep the ferritin levels in patients requiring maintenance therapy below 50 microg/L, with minimally half the number of treatment procedures when compared to current standard therapy by P.

DETAILED DESCRIPTION:
The research population exists of patients with HH ( by genetic analysis confirmed as homozygous for C282Y) living in south-east of the Netherlands and currently treated with phlebotomy as maintenance treatment to keep their serum ferritin levels < 50 ug/l. Ferritin level at start of the inclusion between 30-50ug/l. Exclusion criteria are: patient receiving other therapies such as chelating therapy or forced dietary regimen, further patients with excessive overweight (BMI>35). After enrollment the patients will be randomized to start either with TE or continue with P. After a year of treatment and being at a serum ferritin level <50ug/l, patients will continue the study but then being treated with the other of the two treatments. Randomization will be done by blocked randomization.

ELIGIBILITY:
Inclusion Criteria:

* homozygous for C282Y
* currently treated with phlebotomy as maintenance therapy for at least 6 month
* ferritin level between 30-50 micog/L
* age 18 years an older
* weight more than 50 kg
* signed informed consent
* willingness to fill out additional questionnaires at three points in time

Exclusion Criteria:

* chelating therapy
* forced dietary regime
* aged below 18 years
* excessive overweight ( BMI more than 35)
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The difference in number of required treatments and the interval between treatments per year to keep the serum ferritin levels between 30-50 microg/L | one year after first phlebotomy treatment and one year after first erythrocytapheresis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rombout, MD, Principal Investigator — Sanquin Blood Supply
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands